CLINICAL TRIAL: NCT00993083
Title: A Phase IIA Study to Assess the Safety and Efficacy of a New Influenza Candidate Vaccine MVA-NP+M1 In Healthy Adults
Brief Title: A Study to Assess the Safety and Efficacy of a New Influenza Candidate Vaccine MVA-NP+M1 In Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Professor Adrian Hill, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Flu002
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-01

CONDITIONS: Influenza
Keywords: Influenza; Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccinated (Experimental): 14 volunteers (2 in lead safety group and 12 in main study group) to receive MVA-NP+M1 via the IM route. Volunteers will then be challenged with Influenza 30 days post vaccination.
  Interventions: Biological: MVA-NP+M1
- Control (No Intervention): 12 volunteers who will not receive vaccine but will also be challenged with Influenza on day 30

INTERVENTIONS:
Biological: MVA-NP+M1 — Intramuscular injection at 1.5 x 10^8 pfu/ml at day 0
  Arms: Vaccinated

SUMMARY:
This is a Phase IIa open label, non placebo controlled, non-randomised controlled challenge study. The primary objective of this study is to assess the safety of a new influenza vaccine, MVA-NP+M1, when administered as a single dose to healthy volunteers.

Initially two volunteers will be vaccinated and challenged with Influenza, followed by vaccination of a further 12 volunteers and an Influenza challenge of those 12 along with 12 non-vaccinated controls.

DETAILED DESCRIPTION:
Antibodies against the external proteins of influenza can prevent the virus from infecting cells and either prevent infection or limit the spread of infection. However the surface proteins are highly variable and there is little antibody cross-reactivity between variants. Once a cell has been infected with the virus, it is then vulnerable to T cell attack resulting in the destruction of infected cells so that no more virus can be produced and the infection is controlled. There is evidence from clinical trials of influenza challenge, and animal models that T cell responses can protect in the absence of antibodies. Additionally, since T cells can recognise the highly conserved internal proteins of influenza, cross-subtype protection can be achieved.

Seasonal influenza infection results in a T cell response to the virus which can protect against subsequent infection. However over the course of a few years these responses decline below protective levels. The new vaccine being tested in this study is designed to boost these T cell responses back to protective levels. Even responses that may be too low to be reliably quantified by currently available assays may still be boosted to high levels by a single dose of recombinant MVA. Since the internal proteins vary little between influenza subtypes, this could result in a 'universal' vaccine against influenza A. If the need to continually reformulate the vaccine in response to mutations in the viral coat proteins can be removed, the universal vaccine could be produced in large amounts and used more widely than the existing seasonal 'flu vaccines, thus protecting the population against currently circulating viruses and new virus types that are at present only found in avian species.

There is very little polymorphism of NP and M1 between influenza A isolates. NP is 92% identical between H3N2 and H1N1 strains, and 91% identical between H3N2 and H5N1 strains. M1 is 95% identical between H3N2 and H1N1 strains, and 93% identical between H3N2 and H5N1 strains. This low level of variation appears to allow strong T cell cross-reactivity.

MVA is a highly attenuated strain of vaccinia virus that is unable to replicate efficiently in human cell lines and most mammalian cells. Viral replication is blocked at a late stage of virion assembly, so, importantly, viral and recombinant protein synthesis is unimpaired. This means that MVA is an efficient single round expression vector, incapable of causing infection in mammals. Replication-deficient recombinant MVA has been seen as an exceptionally safe viral vector. This safety in man is consistent with the avirulence of MVA in animal models, where recombinant MVAs have also been shown to be protectively immunogenic as vaccines against viral diseases and cancer. Importantly for a vaccine which may eventually be used in a large proportion of the population, recombinant MVAs expressing HIV antigens have been shown to be safe and immunogenic in HIV-infected subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females aged 18 - 45 years
2. HI titre of less than 10
3. In general good health determined by a screening evaluation (medical history, physical examination, vital signs electrocardiogram (ECG) and clinical safety laboratory tests). ECG and spirometry will be performed at entry into quarantine rather than at screening visit
4. Females should fulfil the following criteria: (i) not pregnant or breastfeeding for the duration of the study and (ii) agree to use a reliable form of contraception for the duration of the study if sexually active
5. Negative HBsAg, HIV and HCV antibody screen
6. Negative class A drugs of abuse screen
7. Have not been vaccinated for Influenza virus in the current season or had a known influenza virus infection in the current season
8. Give written informed consent to participate
9. Willingness to remain in isolation during the challenge phase of the study and to comply with all study requirements
10. Willing and able to communicate with the Investigator and understand the requirements of the study

Exclusion Criteria:

1. Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use of an IMP during the study period
2. Prior receipt of a recombinant MVA vaccine (vaccinees only)
3. Administration of immunoglobulins and/or any blood products within the three months preceding date of enrolment.
4. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months
5. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products. Any allergy to eggs or egg products
6. Any history of anaphylaxis in reaction to vaccination
7. Current cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
8. Serious current psychiatric condition
9. Any other chronic illness requiring hospital specialist supervision
10. Suspected or known current injecting drug or alcohol abuse (as defined by an alcohol intake of greater than 42 units every week)
11. Any other significant disease, disorder or finding, which, in the opinion of the Investigators, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study.
12. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis (see Table 1. Values outside the stated limits of Table 1 need written comment by a physician if considered clinically insignificant).
13. Venous access inadequate for phlebotomy demands of the study
14. Clinically significant abnormality on ECG
15. History since age 13 of asthma of any aetiology
16. Smokers who are unwilling or unable to desist for the duration of the inpatient challenge component of the study
17. Any anatomic or neurologic abnormality impairing the gag reflex or associated with a risk of aspiration
18. Presence of febrile illness or symptoms of upper respiratory tract infection on the day of vaccination (vaccination would be deferred)
19. Presence of febrile illness or symptoms suggestive of influenza between admission for influenza challenge and administration of the challenge inoculum
20. Use of inhaled, topical or systemic steroids in the six months preceding date of enrolment other than occasional use of cutaneous steroid if considered clinically irrelevant to the study by the Investigator..
21. Donation of blood or blood products within 7 days before study entry or at any time during the study
22. Donation of plasma within 7 days of study entry
23. Anti-'flu antibody titre of 10 or greater

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety of a new Influenza vaccine, MVA-NP+M1, when administered to healthy volunteers | 6 months

SECONDARY OUTCOMES:
Cellular immune response generated by a new influenza vaccine MVA- NP+M1 when administered as a single dose to healthy adults. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, DPhil, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Wellcome Trust Clinical Research Facility, University of Southampton, Southampton, Hampshire
  - Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Churchill Hospital, Oxford, Oxfordshire

REFERENCES:
- [Derived] Lillie PJ, Berthoud TK, Powell TJ, Lambe T, Mullarkey C, Spencer AJ, Hamill M, Peng Y, Blais ME, Duncan CJ, Sheehy SH, Havelock T, Faust SN, Williams RL, Gilbert A, Oxford J, Dong T, Hill AV, Gilbert SC. Preliminary assessment of the efficacy of a T-cell-based influenza vaccine, MVA-NP+M1, in humans. Clin Infect Dis. 2012 Jul;55(1):19-25. doi: 10.1093/cid/cis327. Epub 2012 Mar 22. PMID 22441650